CLINICAL TRIAL: NCT03129230
Title: Yulin Orthopedics Hospital of Chinese and Western Medicine
Brief Title: Free Nonvascularized Fibula Autograft for Tumor-like Lesions in Femoral Neck Using in Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yulin Orthopedics Hospital of Chinese and Western Medicine (Other)
Responsible Party: Principal Investigator, Shanchao Luo, Director, Yulin Orthopedics Hospital of Chinese and Western Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20170301c
Record Dates: First submitted 2017-04-05; First posted 2017-04-26 (Actual); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: Bone Diseases
MeSH Terms: conditions — Bone Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Free nonvascularized fibula autograft (Experimental): Sixteen pediatric patients before epiphyseal closure were treated with free nonvascularized fibula autograft after resections of tumor-like lesions in the femoral neck.
  Interventions: Procedure: free nonvascularized fibula autograft

INTERVENTIONS:
Procedure: free nonvascularized fibula autograft — Sixteen pediatric patients before epiphyseal closure were treated with free nonvascularized fibula autograft after resections of tumor-like lesions in the femoral neck between Aug. 2012 and Sep. 2016. All the patients were given supplementary skeletal traction through supracondyle of femur for 4 weeks to 6 weeks after the resections.

SUMMARY:
This study was to evaluate the safety and efficacy of free nonvascularized fibula autograft in the treatment of the femoral neck tumor-like lesions before epiphyseal closure in pediatric patients, by presenting the clinic-radiological outcome and complications.

ELIGIBILITY:
Inclusion Criteria:

1. This retrospective study included pediatric patients before epiphyseal closure with tumor-like lesions in femoral neck.

Exclusion Criteria:

1. pediatric patients with tumor-like lesions in femoral neck after epiphyseal closure;
2. pediatric patients with benign bone tumors and malignant bone tumors in the femoral neck after epiphyseal closure;
3. adult patients with benign or malignant bone tumors and tumor-like lesions in femoral neck.

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2012-08-01 (Actual); Primary Completion 2016-09-01 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
change of peri-implant bone level from baseline at 7 and 54 months | 7 months to 54 months
  Mean follow-up of all the patients after primary surgery was 24 months, ranged 7 months to 54 months.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Yulin Orthopedics Hospital of Chinese and Western Medicine, Yulin, Guangxi

IPD SHARING:
Plan to Share IPD: No